CLINICAL TRIAL: NCT04621149
Title: A Phase 2 Screening Study of Candidate Non-prescription Treatments for COVID-19: A Patient-driven, Randomized, Factorial Study Evaluating Patient-reported Outcomes (PROFACT-01)
Brief Title: An Outpatient Study Investigating Non-prescription Treatments for COVID-19
Acronym: PROFACT-01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit participants due to decline in COVID-19.
Sponsor: Profact, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Profact-01
Record Dates: First submitted 2020-11-05; First posted 2020-11-09 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — chlorine dioxide; Zinc Acetate; Famotidine; Lactoferrin; Tea

STUDY DESIGN:
Intervention Model Description: This will be a randomized, blinded placebo-controlled study with respect to the active treatment vs placebo, and randomized open-label with respect to non-prescription medicine and supplements.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- placebo (Placebo Comparator): 1 liter of filtered water
  Interventions: Other: placebo
- chlorine dioxide aqueous solution (AS) (Active Comparator): 1 liter of filtered water with AS
  Interventions: Other: chlorine dioxide
- placebo with zinc acetate (ZA) (Active Comparator): 1 liter of filtered water with ZA
  Interventions: Dietary Supplement: zinc acetate; Other: placebo
- AS with ZA (Active Comparator): 1 liter of filtered water with AS and ZA
  Interventions: Other: chlorine dioxide; Dietary Supplement: zinc acetate
- placebo with famotidine, lactoferrin and green tea extract (FLG) (Active Comparator): 1 liter of filtered water with FLG
  Interventions: Drug: Famotidine; Other: placebo; Dietary Supplement: lactoferrin, green tea extract
- AS with FLG (Active Comparator): 1 liter of filtered water with AS and FLG
  Interventions: Other: chlorine dioxide; Drug: Famotidine; Dietary Supplement: lactoferrin, green tea extract
- placebo with ZA and FLG (Active Comparator): 1 liter of filtered water with ZA and FLG
  Interventions: Dietary Supplement: zinc acetate; Drug: Famotidine; Other: placebo; Dietary Supplement: lactoferrin, green tea extract
- AS with ZA and FLG (Active Comparator): 1 liter of filtered water with AS, ZA, and FLG
  Interventions: Other: chlorine dioxide; Dietary Supplement: zinc acetate; Drug: Famotidine; Dietary Supplement: lactoferrin, green tea extract

INTERVENTIONS:
Other: chlorine dioxide — chlorine dioxide is an antimicrobial agent used for a variety of purposes including as a water purification product, a disinfectant on food, etc.
  Arms: AS with FLG; AS with ZA; AS with ZA and FLG; chlorine dioxide aqueous solution (AS)
Dietary Supplement: zinc acetate — zinc acetate lozenges have been suggested to have antiviral properties
  Arms: AS with ZA; AS with ZA and FLG; placebo with ZA and FLG; placebo with zinc acetate (ZA)
Drug: Famotidine — famoitidine is a histamine-2 blocker sold over the counter to reduce stomach acid
  Other Names: Pepcid
  Arms: AS with FLG; AS with ZA and FLG; placebo with ZA and FLG; placebo with famotidine, lactoferrin and green tea extract (FLG)
Other: placebo — filtered water
  Other Names: filtered water
  Arms: placebo; placebo with ZA and FLG; placebo with famotidine, lactoferrin and green tea extract (FLG); placebo with zinc acetate (ZA)
Dietary Supplement: lactoferrin, green tea extract — lactoferrin and green tea extract are dietary supplements
  Arms: AS with FLG; AS with ZA and FLG; placebo with ZA and FLG; placebo with famotidine, lactoferrin and green tea extract (FLG)

SUMMARY:
This is a platform study to investigate the effectiveness of a variety of non-prescription approaches for the treatment of non-hospitalized adults recently tested positive for COVID-19.

DETAILED DESCRIPTION:
This study will screen for the activity of a variety of non-prescription approaches for the treatment of non-hospitalized adults recently diagnosed with COVID-19. This will be a randomized, blinded placebo-controlled study with respect to the active treatment (chlorine dioxide) vs placebo, and randomized open-label with respect to a non-prescription medication (famotidine) and supplements including zinc, EGCG and lactoferrin. Treatment will last for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 20-70
4. Confirmed diagnosis of COVID-19 by positive COVID-19 test. Symptoms of a mild degree such that hospitalization is not required. Within 7 days of symptom onset.
5. Ability to drink at least 1 liter of water daily and be willing to adhere to the study regimen

Exclusion Criteria:

1. COVID-19 symptoms of a severe enough nature that requires hospitalization
2. Pregnancy or lactation
3. Diagnosis of diabetes mellitus
4. currently taking paroxetine or digoxin
5. Individuals with diabetes mellitus

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Reduction in Participant Symptoms of COVID-19 | 3 days
  Symptoms of COVID-19 will be evaluated daily using a visual analogue scale

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 days
  Participants will complete a daily assessment for adverse events
Rate of Hospitalization | 28 days
  Admission to Hospital
Change in Oxygen Saturation | 8 days
  Oxygen saturation
Change in Body Temperature | 8 days
  Body temperature

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Murphy, MD, MD(H), Principal Investigator — Profact, Inc.
Locations (1):
- AZ Good Health Center, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343